CLINICAL TRIAL: NCT01522456
Title: Split-face Tolerability Comparison Between Epiduo® (Adapalene and Benzoyl Peroxide) Gel 0.1%/2.5% Versus Retin-A Micro® (Tretinoin Gel) Microsphere, 0.1% in Subjects With Acne Vulgaris
Brief Title: Split-face Tolerability Comparison Between Adapalene-Benzoyl Peroxide Gel Versus Tretinoin Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US10201
Record Dates: First submitted 2012-01-23; First posted 2012-01-31 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2015-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epiduo Gel (Active Comparator): Adapalene 0.1% and benzoyl peroxide 2.5% gel
  Interventions: Drug: Epiduo Gel
- Retin-A Micro Microsphere 0.1% (Active Comparator): Tretinoin gel, 0.1%
  Interventions: Drug: Retin-A Micro Microsphere 0.1%

INTERVENTIONS:
Drug: Epiduo Gel — Once-daily application of fixed dose of adapalene 0.1% and benzoyl peroxide 2.5% in an aqueous based gel.
  Arms: Epiduo Gel
Drug: Retin-A Micro Microsphere 0.1% — Once-daily application of tretinoin gel, 0.1% by weight, in a formulation of porous microspheres in an aqueous gel.
  Arms: Retin-A Micro Microsphere 0.1%

SUMMARY:
To compare the tolerability of Epiduo® (adapalene and benzoyl peroxide) Gel 0.1%/2.5% to Retin-A Micro® (tretinoin gel) microsphere when used by subjects with acne vulgaris for 3 weeks in terms of local tolerability parameters (erythema, dryness, scaling, stinging/burning) and preference.

DETAILED DESCRIPTION:
Adult subjects with acne vulgaris will receive tretinoin gel 0.1% on one side of the face and adapalene 0.1% / benzoyl peroxide 2.5% gel on the other side of the face once daily for a period 3 weeks (22 days). Tolerability assessments (erythema, dryness, scaling, stinging/burning)on both sides of the face will be taken on each visit, on each weekday from from baseline to day 22. The investigator and subjects will respond to user preference questions on days 5, 12, 19, and 22.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of any race
* Subjects 18 years or older
* Subjects with acne vulgaris

Exclusion Criteria:

* Subjects with an allergy to a component of the study drugs (refer to the package inserts for Epiduo Gel and Retin-A Micro 0.1%)
* Subjects with a washout period for topical treatment (less than 1 week for corticosteroids or 4 weeks for retinoids)
* Subjects with a washout period for systemic treatment (less than 1 week for medications that may have increased photosensitivity or 4 weeks for corticosteroids or 24 weeks for oral retinoids)
* Subjects with a sunburn, eczema, atopic dermatitis, perioral dermatitis, rosacea, or other topical conditions on the treatment area
* Subjects with planned unprotected and intense UV exposure during the study (mountain sports, UV radiation, sunbathing, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- Stephens and Associates, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Participants: All subjects randomized into the trial who received Epiduo Gel and Retin-A Micro 0.1% gel on each side of the face
Period: Overall Study
Arm/Group | Total Participants
Started | 73
Completed | 65
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Pregnancy | 1
Not completed — Tolerability Assessment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Total Participants
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Worst Postbaseline Tolerability (Erythema)
Description: Worst postbaseline tolerability assessment for erythema.
Time Frame: Day 1 - Day 22
Population: Safety population
Measure: Number; unit: participants
Groups:
- Epiduo Gel: Fixed dose of adapalene 0.1% and benzoyl peroxide 2.5% gel
  Epiduo Gel : Fixed dose of adapalene 0.1% and benzoyl peroxide 2.5% in an aqueous based gel.
- Retin-A Micro Microsphere 0.1%: Tretinoin gel, 0.1%
  Retin-A Micro Microsphere 0.1% : Tretinoin gel, 0.1% by weight, in a formulation of porous microspheres in an aqueous gel.
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  None | 25 | 28
  Mild | 27 | 24
  Moderate | 19 | 19
  Severe | 2 | 2

2. Secondary Outcome: Tolerability at Day 22 (Erythema)
Description: Tolerability assessments at day 22 for erythema
Time Frame: Day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  None | 36 | 38
  Mild | 33 | 28
  Moderate | 0 | 3
  Severe | 0 | 0
  Data Missing | 4 | 4

3. Secondary Outcome: Tolerability at Day 22 (Dryness)
Description: Tolerability assessments at day 22 for dryness
Time Frame: Day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  None | 44 | 40
  Mild | 25 | 29
  Moderate | 0 | 0
  Severe | 0 | 0
  Data Missing | 4 | 4

4. Other Pre Specified Outcome: User Preference Survey (Investigator)
Description: Response from investigator when asked: "Which side of the face appears to be less irritated?" Data collected from available participants.
Time Frame: Day 5, day 12, day 19, and day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  Day 5 (n=69) | 34 | 35
  Day 12 (n=67) | 34 | 33
  Day 19 (n=65) | 37 | 28
  Day 22 (n=72) | 41 | 31

5. Other Pre Specified Outcome: User Preference Survey (Subjects)
Description: Response from subjects when asked: "Which side of the face feels less irritated?" Data collected from available participants on each assessment day.
Time Frame: Day 5, day 12, day 19, and day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  Day 5 (n=69) | 42 | 27
  Day 12 (n=67) | 33 | 34
  Day 19 (n=65) | 36 | 29
  Day 22 (n=72) | 39 | 33

6. Primary Outcome: Worst Postbaseline Tolerability (Scaling)
Description: Worst postbaseline assessment for scaling.
Time Frame: Day 1 - Day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  None | 25 | 18
  Mild | 34 | 43
  Moderate | 14 | 12
  Severe | 0 | 0

7. Primary Outcome: Worst Postbaseline Tolerability (Dryness)
Description: Worst postbaseline tolerability assessments for dryness.
Time Frame: Day 1 - Day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  None | 34 | 28
  Mild | 35 | 41
  Moderate | 4 | 4
  Severe | 0 | 0

8. Secondary Outcome: Tolerability at Day 22 (Scaling)
Description: Tolerability assessments at day 22 for scaling
Time Frame: Day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  None | 54 | 48
  Mild | 12 | 20
  Moderate | 3 | 1
  Severe | 0 | 0
  Data Missing | 4 | 4

9. Primary Outcome: Worst Postbaseline Tolerability (Stinging/Burning)
Description: Worst postbaseline tolerability assessments for stinging/burning
Time Frame: Day 1 - Day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  None | 51 | 57
  Mild | 18 | 14
  Moderate | 3 | 2
  Severe | 1 | 0

10. Secondary Outcome: Tolerability at Day 22 (Stinging/Burning)
Description: Tolerability assessments at day 22 for stinging/burning
Time Frame: Day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  None | 69 | 69
  Mild | 0 | 0
  Moderate | 0 | 0
  Severe | 0 | 0
  Data Missing | 4 | 4

11. Secondary Outcome: Cumulative Tolerability (Erythema)
Description: Cumulative tolerability assessments for erythema. Cumulative tolerability is defined as the sum of the tolerability scores for erythema. Tolerability was assessed on a 4-point categorical scale(0=none, 1=mild, 2=moderate, 3=severe) for all subjects at each visit.
Time Frame: Day 1 - Day 22
Population: Safety population
Measure: Number; unit: scores on a scale
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
scores on a scale
  1 | 26 | 26
  2 | 56 | 52
  3 | 86 | 79
  4 | 122 | 111
  5 | 164 | 149
  8 | 207 | 187
  9 | 244 | 218
  10 | 287 | 250
  11 | 323 | 286
  12 | 370 | 334
  15 | 410 | 368
  16 | 447 | 400
  17 | 483 | 433
  18 | 517 | 464
  19 | 550 | 495
  22 | 583 | 529

12. Secondary Outcome: Cumulative Tolerability (Scaling)
Description: Cumulative tolerability assessments for scaling. Cumulative tolerability is defined as the sum of the tolerability scores for scaling. Tolerability was assessed on a 4-point categorical scale(0=none, 1=mild, 2=moderate, 3=severe) for all subjects at each visit.
Time Frame: Day 1 - Day 22
Population: Safety population
Measure: Number; unit: scores on a scale
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
scores on a scale
  1 | 1 | 0
  2 | 1 | 0
  3 | 5 | 3
  4 | 11 | 9
  5 | 21 | 26
  8 | 44 | 44
  9 | 71 | 71
  10 | 108 | 108
  11 | 141 | 144
  12 | 182 | 190
  15 | 211 | 221
  16 | 228 | 240
  17 | 246 | 260
  18 | 259 | 282
  19 | 277 | 303
  22 | 295 | 325

13. Secondary Outcome: Cumulative Tolerability (Dryness)
Description: Cumulative tolerability assessments for dryness. Cumulative tolerability is defined as the sum of the tolerability scores for dryness. Tolerability was assessed on a 4-point categorical scale(0=none, 1=mild, 2=moderate, 3=severe) for all subjects at each visit.
Time Frame: Day 1 - Day 22
Population: Safety population
Measure: Number; unit: scores on a scale
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
scores on a scale
  1 | 2 | 1
  2 | 3 | 2
  3 | 6 | 2
  4 | 11 | 4
  5 | 18 | 6
  8 | 30 | 11
  9 | 48 | 22
  10 | 73 | 49
  11 | 99 | 76
  12 | 128 | 107
  15 | 152 | 134
  16 | 178 | 162
  17 | 205 | 188
  18 | 231 | 215
  19 | 256 | 242
  22 | 281 | 271

14. Secondary Outcome: Cumulative Tolerability (Stinging/Burning)
Description: Cumulative tolerability assessments for stinging/burning. Cumulative tolerability is defined as the sum of the tolerability scores stinging/burning. Tolerability was assessed on a 4-point categorical scale(0=none, 1=mild, 2=moderate, 3=severe) for all subjects at each visit.
Time Frame: Day 1 - Day 22
Population: Safety population
Measure: Number; unit: scores on a scale
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
scores on a scale
  1 | 0 | 0
  2 | 0 | 1
  3 | 1 | 2
  4 | 4 | 3
  5 | 9 | 6
  8 | 17 | 8
  9 | 29 | 13
  10 | 42 | 20
  11 | 50 | 25
  12 | 60 | 32
  15 | 61 | 33
  16 | 61 | 33
  17 | 61 | 33
  18 | 61 | 33
  19 | 61 | 33
  22 | 61 | 33

15. Secondary Outcome: Cumulative Tolerability (Combined)
Description: Cumulative tolerability assessments for erythema, scaling, dryness, and stinging/burning. Cumulative tolerability is defined as the sum of the tolerability scores for erythema, scaling, dryness, or stinging/burning. Tolerability was assessed on a 4-point categorical scale(0=none, 1=mild, 2=moderate, 3=severe) for all subjects at each visit.
Time Frame: Day 1 - Day 22
Population: Safety population
Measure: Number; unit: scores on a scale
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
scores on a scale
  1 | 29 | 27
  2 | 60 | 55
  3 | 98 | 86
  4 | 148 | 127
  5 | 212 | 187
  8 | 298 | 250
  9 | 392 | 324
  10 | 510 | 427
  11 | 613 | 531
  12 | 740 | 663
  15 | 834 | 756
  16 | 914 | 835
  17 | 995 | 914
  18 | 1068 | 994
  19 | 1144 | 1073
  22 | 1220 | 1158

16. Other Pre Specified Outcome: Overall Tolerability Preference Survey
Description: Overall tolerability preference survey taken by the subjects. Data collected from available subjects on day 22.
Time Frame: Day 22
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1%
Number analyzed (Participants) | 73 | 73
participants
  ____ spread easier (n=71) | 49 | 22
  ____ absorbed quicker into my skin (n=71) | 45 | 26
  ____ had a more pleasant smell (n=71) | 39 | 32
  ____ felt better on my skin (n=71) | 37 | 34
  ____ left smaller amount of residue on skin (n=71) | 50 | 21
  Overall, I prefer ____ (n=71) | 44 | 27

17. Post Hoc Outcome: Fitzpatrick Skin Type Worst Postbaseline Tolerability Assessment (Erythema)
Description: Worst Postbaseline Tolerability Assessment Grouped by Fitzpatrick Skin Type for Erythema. Fitzpatrick skin type is a numerical classification scale for the color of skin from Type 1 to Type VI. Skin type 1 = always burns and never tans (light, pale skin) and skin type VI = never burns, tans very easily, and is deeply pigmented (black, very dark brown to black skin).
Time Frame: Day 1 - Day 22
Population: Safety Population
Measure: Number; unit: participants
Groups:
- Epiduo Gel (Fitzpatrick Skin Types I-III); Epiduo Gel (Fitzpatrick Skin Types IV-VI): Fixed dose of adapalene 0.1% and benzoyl peroxide 2.5% gel
  Epiduo Gel : Fixed dose of adapalene 0.1% and benzoyl peroxide 2.5% in an aqueous based gel.
- Retin-A Micro (Fitzpatrick Skin Types I-III); Retin-A Micro (Fitzpatrick Skin Types IV-VI): Tretinoin gel, 0.1%
  Retin-A Micro Microsphere 0.1% : Tretinoin gel, 0.1% by weight, in a formulation of porous microspheres in an aqueous gel.
Arm/Group | Epiduo Gel (Fitzpatrick Skin Types I-III) | Retin-A Micro (Fitzpatrick Skin Types I-III) | Epiduo Gel (Fitzpatrick Skin Types IV-VI) | Retin-A Micro (Fitzpatrick Skin Types IV-VI)
Number analyzed (Participants) | 41 | 41 | 32 | 32
participants
  None | 5 | 7 | 20 | 21
  Mild | 18 | 17 | 9 | 7
  Moderate | 16 | 15 | 3 | 4
  Severe | 2 | 2 | 0 | 0

18. Post Hoc Outcome: Fitzpatrick Skin Type Worst Postbaseline Tolerability Assessment (Scaling)
Description: Worst Postbaseline Tolerability Assessment Grouped by Fitzpatrick Skin Type for Scaling. Fitzpatrick skin type is a numerical classification scale for the color of skin from Type 1 to Type VI. Skin type 1 = always burns and never tans (light, pale skin) and skin type VI = never burns, tans very easily, and is deeply pigmented (black, very dark brown to black skin).
Time Frame: Day 1 - Day 22
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel (Fitzpatrick Skin Types I-III) | Retin-A Micro (Fitzpatrick Skin Types I-III) | Epiduo Gel (Fitzpatrick Skin Types IV-VI) | Retin-A Micro (Fitzpatrick Skin Types IV-VI)
Number analyzed (Participants) | 41 | 41 | 32 | 32
participants
  None | 13 | 10 | 12 | 8
  Mild | 19 | 22 | 15 | 21
  Moderate | 9 | 9 | 5 | 3

19. Post Hoc Outcome: Fitzpatrick Skin Type Worst Postbaseline Tolerability Assessment (Dryness)
Description: Worst Postbaseline Tolerability Assessment Grouped by Fitzpatrick Skin Type for Dryness. Fitzpatrick skin type is a numerical classification scale for the color of skin from Type 1 to Type VI. Skin type 1 = always burns and never tans (light, pale skin) and skin type VI = never burns, tans very easily, and is deeply pigmented (black, very dark brown to black skin).
Time Frame: Day 1 - Day 22
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel (Fitzpatrick Skin Types I-III) | Retin-A Micro (Fitzpatrick Skin Types I-III) | Epiduo Gel (Fitzpatrick Skin Types IV-VI) | Retin-A Micro (Fitzpatrick Skin Types IV-VI)
Number analyzed (Participants) | 41 | 41 | 32 | 32
participants
  None | 13 | 14 | 21 | 14
  Mild | 26 | 25 | 9 | 16
  Moderate | 2 | 2 | 2 | 2

20. Post Hoc Outcome: Fitzpatrick Skin Type Worst Postbaseline Tolerability Assessment (Stinging/Burning)
Description: Worst Postbaseline Tolerability Assessment Grouped by Fitzpatrick Skin Type for Stinging/Burning. Fitzpatrick skin type is a numerical classification scale for the color of skin from Type 1 to Type VI. Skin type 1 = always burns and never tans (light, pale skin) and skin type VI = never burns, tans very easily, and is deeply pigmented (black, very dark brown to black skin).
Time Frame: Day 1 - Day 22
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Epiduo Gel (Fitzpatrick Skin Types I-III) | Retin-A Micro (Fitzpatrick Skin Types I-III) | Epiduo Gel (Fitzpatrick Skin Types IV-VI) | Retin-A Micro (Fitzpatrick Skin Types IV-VI)
Number analyzed (Participants) | 41 | 41 | 32 | 32
participants
  None | 28 | 29 | 23 | 28
  Mild | 9 | 10 | 9 | 4
  Moderate | 3 | 2 | 0 | 0
  Severe | 1 | 0 | 0 | 0

21. Post Hoc Outcome: Fitzpatrick Skin Type User Preference Survey at Day 22
Description: User Preference Survey at Day 22 (Safety Population) Grouped by Fitzpatrick Skin Type. Fitzpatrick skin type (FST) is a numerical classification scale for the color of skin from Type 1 to Type VI. Skin type 1 = always burns and never tans (light, pale skin) and skin type VI = never burns, tans very easily, and is deeply pigmented (black, very dark brown to black skin). Two subjects did not participate in the User Preference Survey; as a result, 2 subjects were not included in the FST I - III group results below.
Time Frame: Day 22
Measure: Number; unit: participants
Arm/Group | Epiduo Gel (Fitzpatrick Skin Types I-III) | Retin-A Micro (Fitzpatrick Skin Types I-III) | Epiduo Gel (Fitzpatrick Skin Types IV-VI) | Retin-A Micro (Fitzpatrick Skin Types IV-VI)
Number analyzed (Participants) | 39 | 39 | 32 | 32
participants
  Spread more easily | 22 | 17 | 27 | 5
  Absorbed more quickly | 22 | 17 | 23 | 9
  Smelled better | 20 | 19 | 19 | 13
  Felt better | 15 | 24 | 22 | 10
  Left less residue | 25 | 14 | 25 | 7
  Overall | 20 | 19 | 24 | 8

22. Post Hoc Outcome: Fitzpatrick Skin Type Overall Tolerability Preference Survey Results
Description: Overall Tolerability Preference Survey Results at Day 22 (Safety Population) Grouped by Fitzpatrick Skin Type (FST). Data collected from available subjects on day 22. Fitzpatrick skin type is a numerical classification scale for the color of skin from Type 1 to Type VI. Skin type 1 = always burns and never tans (light, pale skin) and skin type VI = never burns, tans very easily, and is deeply pigmented (black, very dark brown to black skin). One subject did not participate in the User Preference Survey; as a result, 1 subject was not included in the FST I - III group results below.
Time Frame: Day 22
Measure: Number; unit: participants
Arm/Group | Epiduo Gel (Fitzpatrick Skin Types I-III) | Retin-A Micro (Fitzpatrick Skin Types I-III) | Epiduo Gel (Fitzpatrick Skin Types IV-VI) | Retin-A Micro (Fitzpatrick Skin Types IV-VI)
Number analyzed (Participants) | 40 | 40 | 32 | 32
participants
  Overall tolerability preference-investigator | 21 | 19 | 20 | 12
  Overall tolerability preference - subject | 21 | 19 | 18 | 14

ADVERSE EVENTS:
Time Frame: Day 1 - Day 22
Groups:
- Non-application Site: Adverse events occurring on non-application sites
Arm/Group | Epiduo Gel | Retin-A Micro Microsphere 0.1% | Non-application Site
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/73 | 1/73
Other Adverse Events (participants affected / at risk) | 16/73 | 16/73 | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epiduo Gel (N=73) | Retin-A Micro Microsphere 0.1% (N=73) | Non-application Site (N=73)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Epileptic seizure not related to study medicines.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epiduo Gel (N=73) | Retin-A Micro Microsphere 0.1% (N=73) | Non-application Site (N=73)
Dry Skin (Skin and subcutaneous tissue disorders) | 14 (14) | 15 (15) | 0 (0)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less